CLINICAL TRIAL: NCT06261099
Title: The Effect of Telerehabilitation-Based Early Upper Extremity Training on Upper Extremity Function and Proprioception in Stroke Patients
Brief Title: Telerehabilitation-Based Early Upper Extremity Training in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Güler ERTUĞRUL, MSc student, physiotherapist, Suleyman Demirel University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 037
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Stroke, Acute
Keywords: telerehabilitation; Upper Extremity; rehabilitation; Proprioception
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: prospective double-blind, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sealed envelopes will be prepared in advance for randomization and will be marked with numbers 1 and 2, indicating whether they are a study group or a control group. Randomization will be done by a third party unaware of the study content. Randomization order tracking will be done with sequentially numbered containers. Patients participating in the study will be blinded to which treatment group they will be included in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Exercises including upper extremity positioning, overhead activity training, reaching activities, weight transfer exercises, proprioceptive exercises, and daily living activities training will be applied to this group, 5 sessions per week for 6 weeks. Since the functional recovery of the upper extremity after stroke will be slow, the exercise program is planned to be 5 days a week due to the necessity of applying an intense exercise program in the early period. All patients will be asked to perform exercises under the supervision of a physiotherapist as a home program on other days of the week.
- kontrol+ working group (Experimental): Upper extremity positioning, overhead activity training, reaching activities, weight transfer exercises, proprioceptive exercises, and daily living activities training will be applied to this group using the telerehabilitation method, which was applied to the control group in 5 sessions per week for 6 weeks. The telerehabilitation program will be carried out using an application that provides remote video access called Zoom. Since the functional recovery of the upper extremity after stroke will be slow, the exercise program is planned to be 5 days a week due to the necessity of applying an intense exercise program in the early period. All patients will be asked to perform exercises under the supervision of a physiotherapist as a home program on other days of the week.
  Interventions: Other: control + working group

INTERVENTIONS:
Other: control + working group — Upper extremity positioning, overhead activity training, reaching activities, weight transfer exercises, proprioceptive exercises, and daily living activities training will be applied to this group using the telerehabilitation method, which was applied to in 5 sessions per week for 6 weeks.
  Arms: kontrol+ working group

SUMMARY:
Telerehabilitation method, which is an alternative to face-to-face rehabilitation practices for stroke patients who need intensive, regular and long-term rehabilitation in the early period, has been popularly used in recent years. Telerehabilitation is a practice in which the patient participates in the treatment via digital media without the need for the patient to come to the clinic.

DETAILED DESCRIPTION:
After the sociodemographic data of the participants are recorded, Mini Mental Test (MMT) will be applied to evaluate the cognitive status. Upper extremity functions of patients eligible for the study will be evaluated with the Fugl-Meyer Upper Extremity Scale (FM-UE), proprioception evaluation will be evaluated with the Laser-pointer Assisted Angle Reproduction Test, activities of daily living will be evaluated with the Modified Barthel Index, and reaching performance will be evaluated with the Reaching Performance Scale. Characteristics of the patients participating in the study and all outcome measurements before and after treatment will be evaluated by a blinded physiotherapist. A researcher blinded to the exercise groups and evaluation results will perform the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 30-65, with a history of stroke within the last month,
* Mini Mental Score ≥ 24, 1-10 after discharge. on the day,
* patients who can sit for at least 30 seconds, exhibit a hemiparetic condition, and are clinically stable

Exclusion Criteria:

* Flaccid hemiplegia detected by anamnesis and physical examination,
* Has spasticity in the upper extremity with a severity greater than 1+ according to the Modified Ashworth Scale,
* patients with severe dementia and dysfunction of the upper extremity joints due to a previous musculoskeletal disease

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-02-27 (Estimated); Study Completion 2025-11-27 (Estimated)

PRIMARY OUTCOMES:
Mini Mental Test | six weeks
  It is used to evaluate the cognitive status of patients. It is a simple, short and valid test that is widely used in people with stroke. With this test, various cognitive functions of people such as orientation, recording memory, attention and calculation, recall and language are evaluated. The maximum score that can be obtained is 30. Getting a score of 24 or above indicates that the patient's cognitive functions are within normal limits.
Fugl Meyer Motor Function Scale | six weeks
  Motor performance is evaluated in stroke patients. Each item is given a score from 0 to 2, depending on performance: 2 points; complete detailing, 1 point; partial work of details, 0 points; It is given if details cannot be achieved. The maximum motor performance score for the upper extremity is 66 points.
Laser-pointer Assisted Angle Reproduction Test | six weeks
  It evaluates proprioceptive deviation in stroke patients. Shoulder flexion is measured three times at 45◦, 60◦ and 90◦, and upper extremity proprioception is evaluated by taking the average result of the three measurements.
Modified Barthel Index | six weeks
  Determines the functional adequacy, dependency level and rehabilitation services of stroke patients. Items on the scale are rated between 0 and 15 points in 5-point increments depending on the question. 0-20 points are considered fully dependent, 21-61 points are considered highly dependent, 62-90 points are considered moderately dependent, 91-99 points are considered mildly dependent, and 100 points are considered fully independent.
Reaching Performance Scale | six weeks
  It evaluates compensatory movements for upper extremity extension in stroke patients. Scores on items 1 to 5 are used to identify deficiencies in specific aspects of movement, with scores ranging from 0 to 18 being obtained depending on changing performance.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Güler Ertuğrul, Kocaeli, İ̇zmi̇t
  - Suleyman Demirel University, Isparta, Merkez

IPD SHARING:
Plan to Share IPD: No